CLINICAL TRIAL: NCT00721474
Title: An Open-Label, Randomized, Single-Dose, 2-Period Crossover Study to Determine the Effect of a High-Fat Meal on the Relative Bioavailability and Pharmacokinetics of a Single Dose of Bosutinib Administered Orally to Healthy Subjects
Brief Title: Study to Determine the Effect of a High-Fat Meal on the Relative Bioavailability and Pharmacokinetics of a Single Dose of Bosutinib Administered Orally to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3160A4-1110
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Bosutinib fasting
  Interventions: Drug: Bosutinib
- 2 (Experimental): Bosutinib fed
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — Bosutinib fasting
  Arms: 1
Drug: Bosutinib — Bosutinib fed
  Arms: 2

SUMMARY:
A Study to determine if a high-fat meal has an effect on the pharmacokinetics of bosutinib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men, age 18-50;
* Healthy women of nonchildbearing potential, age 18-50.

Exclusion Criteria:

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (plasma concentrations) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tacoma, Washington, United States